CLINICAL TRIAL: NCT05528939
Title: FAACTS: Feasibility/Acceptability of Attentional-Control Training in Survivors
Brief Title: Feasibility/Acceptability of Attentional-Control Training in Survivors
Acronym: FAACTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's National Research Institute (Other)
Collaborators: St. Jude Children's Research Hospital (Other); Children's Hospital of Philadelphia (Other); George Washington University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven J. Hardy, Principal Investigator, Children's National Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00000150; R21CA261877 (NIH)
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Pediatric Cancer; Pediatric ALL; Pediatric Brain Tumor; Attention Difficulties; Cognitive Deficit in Attention
MeSH Terms: conditions — Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Single-blind, randomized, active-control trial using a 1:1 randomization (stratified by diagnosis) to the intervention or a comparison digital activity.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- EndeavorRx (Experimental): Children will be asked to begin digital attentional control training at home within 6 weeks of baseline testing and to complete 6 training missions per day (25-30 minutes), 5 days per week, for 4 weeks (total = 120 training missions).
  Interventions: Device: EndeavorRx
- Control (Active Comparator): An active control program designed to replicate aspects of the intervention (e.g., regular use of digital device to access fun educational activities) while engaging cognitive skills not particularly involving attention.
  Interventions: Other: Control video game

INTERVENTIONS:
Device: EndeavorRx — EndeavorRx is a digital intervention delivered through an action video game that is indicated to improve attention function. EndeavorRx users first complete two discrete tasks: 1) a perceptual discrimination/attention task in which users respond to target stimuli and ignore distractor stimuli (e.g., tapping the screen quickly only when red aliens appear) and 2) a sensorimotor navigation task in which users tilt their device to steer a hovercraft down a river while targeting or avoiding certain objects. Users are subsequently presented with a multitask training session where they complete the perceptual discrimination/attention task and the sensorimotor navigation task simultaneously. Algorithms adapt the program in both real-time and between sessions to automatically adjust the difficulty level.
  Arms: EndeavorRx
Other: Control video game — The active control program, used in previous studies of this intervention, was designed to match EndeavorRx on expectancy, engagement, and time on task in the form of a challenging and engaging digital word game, targeting cognitive domains not targeted by EndeavorRx and not primarily associated with attentional difficulties. Users are instructed to find and connect letters on a grid to spell words; points are awarded based on number of words formed, word length, and the use of unusual letters. There is progression in difficulty to maintain engagement and expectation of benefit from patients and their caregivers.
  Arms: Control

SUMMARY:
This is a multicenter pilot randomized controlled trial, with an active control condition, of the feasibility, acceptability, and preliminary efficacy of EndeavorRx in a cohort of survivors of acute lymphoblastic leukemia or brain tumor ages 8-16 who are > 1 year from the end of therapy.

DETAILED DESCRIPTION:
Survival rates are increasing for common pediatric cancers, including acute lymphoblastic leukemia (ALL) and brain tumors; yet, the life-saving treatments for these cancers place survivors at heightened risk for sustained cognitive effects. Longitudinal research has shown that the cognitive burden of ALL and pediatric brain tumors often consists of impairments in attention, working memory, and executive functioning, which can result in long-term disruption to daily living, socialization, academic achievement, and quality of life. Few non-pharmacological interventions exist to ameliorate these cognitive late effects. EndeavorRx, an FDA-approved electronic attentional-control training program, may be one intervention to help remediate executive functioning difficulties experienced by survivors. Although the program has been efficacious for youth with Attention-Deficit/Hyperactivity Disorder (ADHD), it has not yet been tested among survivors of childhood ALL or brain tumor. We propose to assess the feasibility, acceptability, and preliminary efficacy of EndeavorRx in a pilot randomized, controlled trial. Survivors of ALL or brain tumor who are between the ages of 8 and 16 and have been off-therapy for at least one year will be included. The goal is to enroll and screen approximately 50 survivors across three pediatric oncology centers, in order to identify 40 participants with attention difficulties who will be randomized to one of two treatment arms. Participants will be assigned to either the EndeavorRx intervention, which includes 25-30 minute sessions per day, 5 days per week, for one month, or an active control condition of the same duration and intensity. Patients will undergo neurocognitive testing pre- and post-intervention, and parents will complete questionnaires regarding their child's functioning. It is hypothesized that this attentional-control training program will be both acceptable and feasible, with sufficient enrollment, positive satisfaction ratings, and acceptable treatment adherence. It is also anticipated that participants will show increases in performance-based and parent-rated attention, as compared to those in the active control condition.

ELIGIBILITY:
Inclusion Criteria:

* Aged 8-16 years at time of screening.
* History of diagnosis of acute lymphoblastic leukemia (ALL) or brain tumor (BT).
* At least 1 year from completion of planned therapy and stable from a disease standpoint.
* Participating child and caregiver are fluent in spoken English.
* Availability of a caregiver who is willing and capable of providing support and supervision during cognitive training.
* Participating child is either not taking any prescribed stimulant medication for attention difficulties or has been prescribed a stable dose of stimulant medication for attention difficulties for at least 30 days prior to enrollment.
* Only patients with a T-score ≥ 75th percentile on the CPT-3 Omission Errors scale or on the BRIEF-2 Cognitive Regulation Index will be randomized.

Exclusion Criteria:

* A history of photosensitive seizures.
* A motor, visual, or auditory handicap that prevents computer use.
* A mental health condition that precludes, or takes treatment precedence over, participation in the cognitive training.
* Participants identified during the baseline assessment as having a full-scale IQ < 80, as estimated by WASI-II (Vocabulary and Matrix Reasoning), will not be randomized.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-06-14 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility assessed by patient/family interest | Baseline
  Feasibility will be determined by examining the proportion of eligible patients/families approached about the study who enroll
Feasibility assessed by EndeavorRx training adherence rates | After completion of 4 weeks of EndeavorRx training
  Participants will be asked to complete 6 EndeavorRx training missions per day, 5 days per week, for 4 weeks, resulting in a possible training of 120 missions. Feasibility will be evaluated by examining the proportion of the sample that completes at least 60 EndeavorRx missions (50%).
Feasibility assessed by reports of technical ease-of-use and satisfaction | End of training (+4 weeks)
  Children and caregivers will be asked, "How easy or difficult was it to access (e.g., turn on device, start the program, use the program)" using a 5-point Likert scale (5 = "Very Easy"). Families will also be asked, "How satisfied or unsatisfied are you with your experience using EndeavorRx?" using a 5-point Likert scale (5 = "Very Satisfied").

SECONDARY OUTCOMES:
Change from baseline inattention assessed by Omission Errors on the Conners' Continuous Performance Test, 3rd Edition (CPT-3) at end of training | Baseline and end of training (+4 weeks)
  The Conners CPT-3 is a standardized computer-administered assessment that uses T scores (M=50, SD=10) where higher scores indicate greater attention problems
Change from baseline inattention assessed by Omission Errors on the Conners' Continuous Performance Test, 3rd Edition (CPT-3) at 4-month follow-up (16 weeks post-training/control +/- 4 weeks) | Baseline and 4 months after end of training (16 weeks post-training/control +/- 4 weeks)
  The Conners CPT-3 is a standardized computer-administered assessment that uses T scores (M=50, SD=10) where higher scores indicate greater attention problems
Change from baseline inattention assessed by the ADHD Rating Scale, Fifth Edition (ADHD-RS-5) Inattention subscale at end of training | Baseline and end of training (+4 weeks)
  The ADHD-RS-5 is a caregiver-reported questionnaire measure of attentional symptoms based on DSM-5 criteria where higher raw scores indicate greater attention problems
Change from baseline inattention assessed by the ADHD Rating Scale, Fifth Edition (ADHD-RS-5) Inattention subscale at 4-month follow-up (16 weeks post-training/control +/- 4 weeks) | Baseline and 4 months after end of training (16 weeks post-training/control +/- 4 weeks)
  The ADHD-RS-5 is a caregiver-reported questionnaire measure of attentional symptoms based on DSM-5 criteria where higher raw scores indicate greater attention problems
Change from baseline inhibitory control assessed by the Behavior Rating Inventory of Executive Functioning, Second Edition (BRIEF-2) Inhibit subscale at end of training | Baseline and end of training (+4 weeks)
  The BRIEF-2 is a caregiver-reported questionnaire measure of executive functioning that uses T scores (M=50, SD=10) where higher scores indicate greater problems with executive functioning
Change from baseline inhibitory control assessed by the Behavior Rating Inventory of Executive Functioning, Second Edition (BRIEF-2) Inhibit subscale at 4-month follow-up (16 weeks post-training/control +/- 4 weeks) | Baseline and 4 months after end of training (16 weeks post-training/control +/- 4 weeks)
  The BRIEF-2 is a caregiver-reported questionnaire measure of executive functioning that uses T scores (M=50, SD=10) where higher scores indicate greater problems with executive functioning
Change from baseline executive functioning assessed by the Behavior Rating Inventory of Executive Functioning, Second Edition (BRIEF-2) Cognitive Regulation Index (CRI) at end of training | Baseline and end of training (+4 weeks)
  The BRIEF-2 is a caregiver-reported questionnaire measure of executive functioning that uses T scores (M=50, SD=10) where higher scores indicate greater problems with executive functioning
Change from baseline executive functioning assessed by the Behavior Rating Inventory of Executive Functioning, Second Edition (BRIEF-2) Cognitive Regulation Index (CRI) at end of training | Baseline and 4 months after end of training (16 weeks post-training/control +/- 4 weeks)
  The BRIEF-2 is a caregiver-reported questionnaire measure of executive functioning that uses T scores (M=50, SD=10) where higher scores indicate greater problems with executive functioning

CONTACTS AND LOCATIONS:
Overall Officials: Steven Hardy, Ph.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No